CLINICAL TRIAL: NCT03583008
Title: Supporting Use of AC Through Provider Profiling of Oral AC Therapy for AF
Acronym: SUPPORT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Alok Kapoor, Assistant Professor, University of Massachusetts Medical School, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00012403
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; Prescribing Practices; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation (AC) Intervention (Experimental): Providers in this arm will receive supportive tools including Anticoagulation (AC) Intervention--Prescribing Practices and Anticoagulation (AC) Intervention--Academic Detailing to help them assess their Anticoagulant (AC) prescribing practices and will also meet with the study investigators for academic detailing.
  Interventions: Behavioral: Anticoagulation (AC) Intervention--Academic Detailing; Behavioral: Anticoagulation (AC) Intervention--Prescribing Practices
- Control (No Intervention): Providers in this arm will not receive any intervention.

INTERVENTIONS:
Behavioral: Anticoagulation (AC) Intervention--Academic Detailing — One hour online web-based academic detailing session to develop an anticoagulant (AC) learning plan.
  Arms: Anticoagulation (AC) Intervention
Behavioral: Anticoagulation (AC) Intervention--Prescribing Practices — Education and support related to anticoagulant prescribing practices.
  Arms: Anticoagulation (AC) Intervention

SUMMARY:
The SUPPORT-AF study aims to improve rates of anticoagulation (AC) in atrial fibrillation (AF) patients by developing and delivering supportive tools and educational materials to providers treating patients with AF. The investigators hypothesize that AC percentage will increase among providers receiving tools and educational content.

DETAILED DESCRIPTION:
Nearly 1 million patients with atrial fibrillation (AF) who meet guideline criteria for anticoagulation (AC) are being left untreated, often due to providers over-estimating risks of bleeding and falling and under-estimating risks of stroke. The objective of this project is to improve rates of adherence to AC guidelines by creating supportive and educational materials for cardiology as well as primary care providers to evaluate the risks and benefits of prescribing AC to patients with AF. The investigators will email providers individual auto-updating reports containing their AC prescription rate compared to their peers and compared to practice level AC prescription goal. This report will also contain a list of the provider's AF patients who are eligible to receive AC based on their CHA2DS2-VASc stroke risk score ≥ 2 and a list of eligible AF patients with upcoming appointments to focus providers on an actionable group of patients with whom they might review the use of AC. The investigators will also message providers through the EHR prior to an upcoming appointment with an eligible patient reminding them to discuss AC if they deem appropriate. In addition, the investigators will directly engage with providers through academic teledetailing to educate providers on AC and address misconceptions and barriers to initiating or resuming AC in AF patients.

ELIGIBILITY:
Inclusion Criteria:

* University of Massachusetts providers caring for patients aged 18 years and older with ICD-10 diagnostic code consistent with AF or atrial flutter who had a visit with a primary care provider or
* cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the electronic medical record (EHR).

Exclusion Criteria:

* University of Massachusetts providers who do not care for patients aged 18 years and older with ICD-10 diagnostic code consistent with AF or atrial flutter who had a visit with a primary care provider or
* cardiovascular medicine specialist in the previous one year with the diagnosis of AF present as an active diagnosis in the EHR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change to Provider prescription rates | Intervention to three months post intervention.
  The first primary outcome measure is to determine the impact of the intervention on provider prescribing rates (increase, decrease, same)
Change to Individual patient Anticoagulation (AC) status | Intervention to three months post intervention.
  The effect of the intervention on individual patient anti-coagulation status as demonstrated by random effects logistic regression models for post-intervention AC status (anticoagulated / not anticoagulated) as a function of pre-intervention AC status.

SECONDARY OUTCOMES:
Change in provider confidence in applying evidence to balance stroke prevention with harm. | Intervention to three months post intervention.
  The change in provide confidence as assessed by confidence questions included in the provider survey distributed with the AC Provider Profile. More specifically, the change is calculated with an average score for each item in the confidence survey, using a four-point scale based on four response choices - not confident through very confident.

CONTACTS AND LOCATIONS:
Overall Officials: Alok Kapoor, MD, MSca, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapoor A, Amroze A, Vakil F, Crawford S, Der J, Mathew J, Alper E, Yogaratnam D, Javed S, Elhag R, Lin A, Narayanan S, Bartlett D, Nagy A, Shagoury BK, Fischer MA, Mazor KM, Saczynski JS, Ashburner JM, Lopes R, McManus DD. SUPPORT-AF II: Supporting Use of Anticoagulants Through Provider Profiling of Oral Anticoagulant Therapy for Atrial Fibrillation: A Cluster-Randomized Study of Electronic Profiling and Messaging Combined With Academic Detailing for Providers Making Decisions About Anticoagulation in Patients With Atrial Fibrillation. Circ Cardiovasc Qual Outcomes. 2020 Feb;13(2):e005871. doi: 10.1161/CIRCOUTCOMES.119.005871. Epub 2020 Feb 17. PMID 32063041